CLINICAL TRIAL: NCT05955222
Title: Clinical Performance Comparison of Different Occlusal Splint Materials: a Clinical Study
Brief Title: Clinical Performance of CAD/CAM Splint Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Bilge Gokcen-Rohlig, Professor Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDK-2020-35910
Record Dates: First submitted 2023-07-01; First posted 2023-07-21 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: TMD
Keywords: occlusal splint; CAD/CAM splint; clinical performance
MeSH Terms: interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: The study is designed as a prospective, randomized, double-blind in-vivo study
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will not know which group they are assigned. Also the clinician who is going to make the examinations before and after the study will not be aware of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PEEK splint group (Experimental): Patients received splints produced from PEEK blocks
  Interventions: Device: PEEK
- PMMA splint group (Experimental): Patients received splints produced from PMMA blocks
  Interventions: Device: PMMA
- Traditional splint group (Active Comparator): Patients received splints produced fabricated traditional methods (vacuum forming )
  Interventions: Device: Traditional

INTERVENTIONS:
Device: PEEK — Participants receiving splints produced with CAD/CAM from PEEK blocks,
  Other Names: bite splints
  Arms: PEEK splint group
Device: PMMA — Participants receiving splints produced with CAD/CAM from PMMA blocks,
  Other Names: PMMA splints
  Arms: PMMA splint group
Device: Traditional — Participants receiving splints from vacuum forming system
  Other Names: traditional splints
  Arms: Traditional splint group

SUMMARY:
The goal of this clinical study is to compare the performance of computer aided designed and computer aided manufactured (CAD/CAM) occlusal splints with splints produced with conventional methods. The main questions this clinical study aims to answer are:

* Do CAD/CAM splints have the same therapeutic effect as the traditional splints ?
* Do CAD/CAM splints demonstrate better surface wear and fit and lower wear in opposing jaw than traditional splints ?
* Is objective pain evaluation of the patient better with CAD/CAM splints ?

Participants were asked to use the splints for 6 months, 8 hours a day and come for follow-up appointments 3 times during this 6 month period:

* Delivery appointment
* First appointment: one week later after delivery appointment
* Last appointment: 6 months after delivery appointment Researchers compared CAD/CAM groups with traditional group to see the clinical performance of the CAD/CAM groups.

DETAILED DESCRIPTION:
24 patients applying to Istanbul University Faculty of Dentistry Department of Prosthodontics and diagnosed with Diagnostic Criteria/ Temporomandibular Disorders (DC/TMD) protocol were included in the study. The patients were randomly divided into 3 groups (n=8); PEEK group (PEEKG), PMMA group (PMMAG), and control group (CG). Dental stone casts of the upper and the lower jaws of the patients were obtained by condensation type silicone impression material and occlusal splints were fabricated in study groups with digital method (designed and milled, manufactured with CAD/CAM) either from PEEK blocks or PMMA blocks and in control group with traditional vacuum pressing machine and adapted by the clinician at chairside. The patients wore the splints for 6 months. Surface roughness, surface wear, fit of the splints and patient satisfaction as well as therapeutic effect of the splints were examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with TMD according to DC/TMD
* Aged between 18 and 65

Exclusion Criteria:

* Patients with removable dentures
* Patients diagnosed with Disc displacement without reduction according to DC/TMD
* Patients receiving medication for psychological disorders
* Patients diagnosed with systemic joint disorders
* Pregnant
* Patients who has received TMD treatment in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Measurement of occlusal surface change | Baseline and 6 months
  Amount of material loss on the occlusal surface of the splints were determined by superimposition of the scannings which were obtained at the base line and at the end of the study. The surfaces were scanned with a professional reference scanner (Solutionix C500 Optical 3D Measuring System,2018,South Korea) and the data obtained were aligned for the best fit algorithm and digital evaluations were performed with the Geomagic Control (2021,USA) software program with an accuracy of 0.001 mm. Surface abrasions were determined by superposition at 24 different predetermined points.
Measurement of the opposing teeth hard tissue change | Baseline and 6 months
  Hard tissue wear on opposing teeth were determined by superimposition of the casts of the patients which were obtained at the base line and at the end of the study. The cast models were scanned with a professional reference scanner (Solutionix C500 Optical 3D Measuring System,2018,South Korea) and the data obtained were aligned for the best fit algorithm. Evaluations were performed with the Geomagic Control (2021,USA) software program with an accuracy of 0.001 mm. Surface abrasions were determined by superposition at 30 different predetermined points.
Evaluation of the Fit of the splint | Baseline
  The cameo surfaces of the splints were scanned for the evaluation of integral accuracy of the splints and superimposed with the Standard Triangle Language (STL) data of dental arch. The maxillary cast models and the cameo surface of the occlusal splints were scanned with a professional reference scanner (Solutionix C500 Optical 3D Measuring System,2018,South Korea) and the data obtained were aligned for the best fit algorithm. Fit evaluations were performed with the Geomagic Control (2021,USA) software program with an accuracy of 0.001 mm. Surface abrasions were determined by superposition at 24 different predetermined points.
Pain change | baseline and 6 months
  Patients were examined according to DC/TMD (Diagnostic Criteria/ Temporomandibular Disorders) protocol and Clinical examination form of the DC/TMD protocol was used. The patients were examined before and after the treatment. The pain scores of masticatory muscles as well as pain during mandibular movements were recorded.
Subjective pain change | baseline and 6 months
  Patient's evaluations of their overall pain were with performed with VAS (Visual analogue scale). VAS scores ranges from 0 to 100 with the leftmost point indicating 'very poor' and the rightmost 'very good'. The patients were asked to report their pain before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Gokcen Rohlig, Prof. Dr., Study Chair — Istanbul University
Locations (1):
- ıstanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No